CLINICAL TRIAL: NCT01274182
Title: A Randomized, Double-blind, Controlled Study to Evaluate PK, PD, Safety and Efficacy of GP2013 and Rituximab in Patients With Rheumatoid Arthritis Refractory or Intolerant to Standard DMARDs and up to Three Anti-TNF Therapies.
Brief Title: GP2013 in the Treatment of RA Patients Refractory to or Intolerant of Standard Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sandoz (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GP13-201; 2010-021184-32 (EudraCT Number); GPN013A2301 (Other: Novartis)
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Results first posted 2018-01-24 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GP2013 (Experimental)
  Interventions: Biological: GP2013
- MabThera (Active Comparator)
  Interventions: Biological: MabThera
- Rituxan (Active Comparator)
  Interventions: Biological: Rituxan

INTERVENTIONS:
Biological: GP2013 — 1000 mg iv infusion on two separate occasions, two weeks apart (i.e. on Day 1 and on Day 15)
  Arms: GP2013
Biological: MabThera — 1000 mg iv infusion on two separate occasions, two weeks apart (i.e. on Day 1 and on Day 15)
  Other Names: EU-Rituximab
  Arms: MabThera
Biological: Rituxan — 1000 mg iv infusion on two separate occasions, two weeks apart (i.e. on Day 1 and on Day 15)
  Other Names: US-Rituximab
  Arms: Rituxan

SUMMARY:
The purpose of this study is to determine the PK/PD, efficacy and safety of GP2013 in patients with severe rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis as defined by the 1987 ACR classification
* Severe active seropositive disease
* Inadequate response or intolerance to other DMARDs and anti-TNFs
* Treatment with Methotrexate

Exclusion Criteria:

* Patients with systemic manifestations of rheumatoid arthritis
* Female patients nursing
* Women of childbearing potential unless using birth control
* Active infection
* Known immunodeficiency syndrome
* Positive Hepatitis B surface antigen or antibodies to Hepatitis C
* History of cancer

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2011-01; Primary Completion 2016-01 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandoz Biopharmaceuticals, Study Director — Sandoz
Locations (57):
- United States (16):
  - Miller Clinical Research, Los Angeles, California
  - Bluegrass Community Research, Inc., Lexington, Kentucky
  - Klein & Associates, Cumberland, Maryland
  - Klein & Associates, Hagerstown, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Innovative Health Research, Las Vegas, Nevada
  - DJL Clinical Research PLLC, Charlotte, North Carolina
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Center of Reading LLC, Wyomissing, Pennsylvania
  - Low Country Rheumatology, PA, Charleston, South Carolina
  - Regional Health Clinical Research, Rapid City, South Dakota
  - West Tennessee Research Institute, Jackson, Tennessee
  - Arthritis & Osteoporosis Center of South Texas, San Antonio, Texas
  - The Seattle Arthritis Center, Seattle, Washington
- Investigative Site, Buenos Aires, Argentina
- Austria (2):
  - Investigative Site, Innsbruck
  - Investigative Site, Vienna
- Belgium (2):
  - Investigative site, Kortrijk
  - Investigative site, Merksem
- Brazil (3):
  - Investigative Site, Curitiba
  - Investigative Site, Goiânia
  - Investigative Site, São Paulo
- North Estonia Medical Centre Foundation, Tallinn, Estonia
- France (5):
  - Investigative Site, Amiens
  - Investigative site, Cahors
  - Investigative Site, Corbeil-Essonnes
  - Investigative site, La Gaillarde
  - Investigative Site, Orléans
- Germany (10):
  - Investigative Site, Frankfurt
  - Investigative Site, Freiburg im Breisgau
  - Investigative Site, Göttingen
  - Investigative Site, Hildesheim
  - Investigative Site, Jena
  - Investigative Site, München
  - Investigative Site, Nuremberg
  - Investigative Site, Ratingen
  - Investigative Site, Regensburg
  - Investigative Site, Würzburg
- Hungary (2):
  - Pest Megyei Flór Ferenc, Kistarcsa
  - Megyei Csolnoky Ferenc Kórház Nonprofit Zrt., Veszprém
- India (6):
  - Investigative site, Ajmer
  - Investigative Site, Bangalore
  - Investigative Site, Hyderabad
  - Investigative Site, Jaipur
  - Investigative Site, New Delhi
  - Investigative Site, Secunderabad
- Investigative Site, Milan, Italy
- Romania (2):
  - Investigative site, Bucharest
  - Investigative site, Cluj-Napoca
- Spain (4):
  - Investigative Site, Madrid
  - Investigative Site, Mérida
  - Investigative site, Santiago de Compostela
  - Investigative Site, Seville
- Turkey (Türkiye) (2):
  - Investigative Site, Istanbul
  - Investigative Site, Izmir

REFERENCES:
- [Derived] Smolen JS, Cohen SB, Tony HP, Scheinberg M, Kivitz A, Balanescu A, Gomez-Reino J, Cen L, Zhu P, Shisha T. A randomised, double-blind trial to demonstrate bioequivalence of GP2013 and reference rituximab combined with methotrexate in patients with active rheumatoid arthritis. Ann Rheum Dis. 2017 Sep;76(9):1598-1602. doi: 10.1136/annrheumdis-2017-211281. Epub 2017 Jun 21. PMID 28637670

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GP2013 | MabThera | Rituxan
Started | 133 | 87 | 92
24 Weeks | 123 | 83 | 84
Completed | 112 | 69 | 80
Not Completed | 21 | 18 | 12
Not completed — Unsatisfactory therapeutic effect | 6 | 3 | 4
Not completed — Adverse Event | 4 | 5 | 3
Not completed — Withdrawal by Subject | 5 | 5 | 3
Not completed — Lost to Follow-up | 2 | 3 | 1
Not completed — Protocol Violation | 3 | 2 | 0
Not completed — Death | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | GP2013 | MabThera | Rituxan | Total
Number analyzed (Participants) | 133 | 87 | 92 | 312
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.42 (11.779) | 52.17 (12.531) | 54.95 (10.750) | 54.10 (11.701)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 73 | 78 | 262
  Male | 22 | 14 | 14 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 12 | 12 | 0 | 24
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 1 | 6 | 6 | 13
  White | 117 | 68 | 75 | 260
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 11 | 13
Region of Enrollment [Number; unit: participants]
  Argentina | 8 | 3 | 9 | 20
  Austria | 7 | 10 | 3 | 20
  Turkey | 4 | 1 | 2 | 7
  Romania | 9 | 8 | 6 | 23
  Belgium | 1 | 4 | 0 | 5
  United States | 10 | 0 | 19 | 29
  Brazil | 19 | 12 | 19 | 50
  Italy | 5 | 3 | 3 | 11
  France | 4 | 1 | 0 | 5
  Germany | 31 | 17 | 14 | 62
  India | 12 | 12 | 0 | 24
  Spain | 13 | 16 | 4 | 33
  Russia | 6 | 0 | 11 | 17
  Hungary | 3 | 0 | 1 | 4
  Estonia | 1 | 0 | 1 | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] — Population: Analysis done on data of BMI available at the baseline visit.
  kg/m2
    number analyzed (Participants) | 133 | 85 | 92 | 310
    (all) | 27.37 (6.230) | 27.25 (6.000) | 29.66 (6.606) | 28.02 (6.353)
Duration of Rheumatoid Arthritis(RA) [Mean (Standard Deviation); unit: years] — Time in years since initial diagnosis of RA Population: Analysis done on data of Duration of RA available at the baseline visit
  years
    number analyzed (Participants) | 133 | 86 | 92 | 311
    (all) | 10.53 (8.074) | 10.81 (7.137) | 11.10 (8.299) | 10.78 (7.874)
Number of patients having received 1, 2 or >2 TNF inhibitor therapies. [Count of Participants; unit: Participants]
  1 | 109 | 70 | 73 | 252
  2 | 18 | 16 | 13 | 47
  >2 | 6 | 1 | 6 | 13
Disease Activity Score 28 joint count - C-reactive proteine (DAS28-CRP) [Mean (Standard Deviation); unit: units on a scale] — In order to calculate the DAS28(CRP) the number of tender joints and swollen joints were assessed using 28-joint count (tender28 and swollen28).The patient's global assessment of disease activity (GH) measured on a Visual Analogue Scale (VAS from 0mm - best to 100mm - worst) was obtained.
  DAS28(CRP) = 0.56 * sqrt(tender28) + 0.28* sqrt(swollen28) + 0.36 * ln(CRP+1) + 0.014 * GH + 0.96 The DAS28(CRP) provides a number on a scale from 0 to 10 indicating the current activity of the RA, while lower values correspond with less disease activity. A decrease in DAS28 signifies a clinical improvement Population: Analysis done on data of DAS28-CRP available at the baseline visit
  units on a scale
    number analyzed (Participants) | 132 | 87 | 91 | 310
    (all) | 5.83 (0.922) | 5.85 (0.880) | 5.91 (1.009) | 5.86 (0.935)
Dose of methotrexate at baseline [Mean (Standard Deviation); unit: mg/week] — Population: Analysis done on data of Methotrexate use available at the baseline visit
  mg/week
    number analyzed (Participants) | 131 | 84 | 91 | 306
    (all) | 15.09 (4.856) | 14.65 (5.154) | 15.29 (4.888) | 15.03 (4.939)
Anti-drug antibodies (ADA) [Count of Participants; unit: Participants]
  Negative | 132 | 85 | 87 | 304
  Positive | 0 | 2 | 3 | 5
  Missing | 1 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: AUC(0-inf) of GP2013, MabThera and Rituxan Following IV Infusion in Patients With RA
Description: Area under the curve AUC(0-inf) calculated based on serum samples, collected from baseline up to 24 weeks: Day 1, 4, 8, 15, 18, 29, 57, 85,113 and 169
Time Frame: From baseline to 24 weeks
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*mcg/mL
Arm/Group | GP2013 | MabThera | Rituxan
Number analyzed (Participants) | 124 | 79 | 80
day*mcg/mL | 7627.44 (38.60) | 6896.97 (40.56) | 7536.89 (40.28)
Statistical Analysis 1: Comparison: GP2013 vs MabThera; PK bioequivalence is defined as AUC(0-inf) of the drugs being comparable, i.e. the two-sided 90% CI for the ratio of the geometric means (GP2013/MabThera) is within the predefined bioequivalence limits of 0.8 to 1.25; Test type: Equivalence — The PK parameters were transformed prior to analysis using a logarithmic transformation. An analysis of variance (ANOVA) was used to analyze the transformed data including treatment group only as a factor in the model. The confidence interval for the difference between the two products on the transformed scale was obtained from the ANOVA model, which was then be back-transformed (exp base e) to obtain the confidence interval for the ratio on the original scale; Geometric mean ratio = 1.106, 90% CI 2-sided [1.010 to 1.210] — GP2013 arm is the numerator and MabThera arm is the denominator
Statistical Analysis 2: Comparison: GP2013 vs Rituxan; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric mean ratio = 1.012, 90% CI 2-sided [0.925 to 1.108] — GP2013 arm is the numerator and Rituxan arm is the denominator
Statistical Analysis 3: Comparison: MabThera vs Rituxan; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric mean ratio = 1.093, 90% CI 2-sided [0.989 to 1.208] — Rituxan arm is the numerator and MabThera arm is the denominator

2. Secondary Outcome: Maximum Serum Concentration (Cmax) of GP2013, MabThera and Rituxan Following IV Infusion in Patients With RA
Description: Maximum serum concentration (Cmax) after the first infusion of GP2013, MabThera and Rituxan in patients with RA. Samples collected from baseline up to 24 weeks: Day 1, 4, 8, 15, 18, 29, 57, 85,113 and 169.
Time Frame: From baseline to week 24
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | GP2013 | MabThera | Rituxan
Number analyzed (Participants) | 120 | 78 | 82
mcg/mL | 361.53 (40.82) | 319.80 (42.75) | 335.88 (42.65)
Statistical Analysis 1: Comparison: GP2013 vs Rituxan; To conclude bioequivalence the 90% CI must be entirely within the standard equivalence limits of 0.8-1.25; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric mean ratio = 1.076, 90% CI 2-sided [0.979 to 1.184] — GP2013 arm is the numerator and Rituxan arm is the denominator
Statistical Analysis 2: Comparison: GP2013 vs MabThera; To conclude bioequivalence the 90% CI must be entirely within the standard equivalence limits of 0.8-1.25; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric mean ratio = 1.131, 90% CI 2-sided [1.027 to 1.244] — GP2013 arm is the numerator and MabThera arm is the denominator
Statistical Analysis 3: Comparison: MabThera vs Rituxan; To conclude bioequivalence the 90% CI must be entirely within the standard equivalence limits of 0.8-1.25; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric mean ratio = 1.050, 90% CI 2-sided [0.946 to 1.167] — Rituxan arm is the numerator and MabThera arm is the denominator

3. Secondary Outcome: Area Under the Effect Curve From Baseline to Day 14 (AUEC(0-14d)) of Percent B-cells of GP2013, MabThera and Rituxan in Patients With RA
Description: Area under the effect curve of percent change of peripheral B-cell count from baseline to Day 14 (AUEC(0-14d)) of GP2013, MabThera and Rituxan in patients with RA
Time Frame: 14 days
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: % * day
Arm/Group | GP2013 | MabThera | Rituxan
Number analyzed (Participants) | 110 | 76 | 80
% * day | 1226.53 (2.83) | 1201.15 (8.91) | 1240.57 (1.95)
Statistical Analysis 1: Comparison: GP2013 vs Rituxan; To conclude equivalence the 95% CI must be entirely within the standard equivalencelimits of 0.8-1.25; Test type: Equivalence — Ratio of geometric means and 95% confidence interval were estimated by an analysis of variance (ANOVA) on log-transformed PD parameter with treatment as the factor. Results were then back-transformed to the original scale; Geometric mean ratio = 0.989, 95% CI 2-sided [0.974 to 1.004] — GP2013 arm is the numerator and Rituxan arm is the denominator
Statistical Analysis 2: Comparison: GP2013 vs MabThera; To conclude equivalence the 95% CI must be entirely within the standard equivalencelimits of 0.8-1.25; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean ratio = 1.021, 95% CI 2-sided [1.003 to 1.040] — GP2013 arm is the numerator and MabThera arm is the denominator
Statistical Analysis 3: Comparison: MabThera vs Rituxan; To conclude equivalence the 95% CI must be entirely within the standard equivalence limits of 0.8-1.25; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean ratio = 1.033, 95% CI 2-sided [1.016 to 1.050] — Rituxan arm is the numerator and MabThera arm is the denominator

4. Secondary Outcome: Change From Baseline in DAS28(CRP) at Week 24
Description: Change from baseline in Disease Activity Score 28 joint count - C-reactive proteine DAS28(CRP) at Week 24.
  In order to calculate the DAS28(CRP) the number of tender joints and swollen joints were assessed using 28-joint count (tender28 and swollen28).The patient's global assessment of disease activity (GH) measured on a Visual Analogue Scale (VAS from 0mm - best to 100mm - worst) was obtained.
  DAS28(CRP) = 0.56 * sqrt(tender28) + 0.28* sqrt(swollen28) + 0.36 * ln(CRP+1) + 0.014 * GH + 0.96 The DAS28(CRP) provides a number on a scale from 0 to 10 indicating the current activity of the RA, while lower values correspond with less disease activity. A decrease in DAS28 signifies a clinical improvement.
Time Frame: 24 weeks
Population: PP analysis set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- GP2013 Part I: This is the subgroup of patients in the GP2013 treatment arm, who were enrolled in the study Part I.
  Efficacy comparisons between GP2013 and MabThera were done in the study Part I on patients enrolled only in the study Part I
Arm/Group | GP2013 | MabThera | Rituxan | GP2013 Part I
Number analyzed (Participants) | 128 | 82 | 85 | 85
units on a scale | -2.07 (0.103) | -2.23 (0.143) | -1.99 (0.126) | -2.16 (0.142)
Statistical Analysis 1: Comparison: GP2013 vs Rituxan; To conclude non-inferiority the upper 95% CI should be less than or equal to 0.6. This margin was statistically justified by the results of the REFLEX (Randomized Evaluation of Long-Term Efficacy of Rituximab in RA) trial (Cohen et al 2006) providing a 95% CI for the mean difference between rituximab/MTX and MTX alone of (-1.74;-1.25). The margin of 0.6 was determined by retaining more than 50% of the reference treatment effect which was considered clinically acceptable; Test type: Non-Inferiority — The non-inferiority margin is further justified by the EULAR criteria which define "no response" as change from baseline being < 0.6. LS means, standard errors and 95% CI were estimated by a repeated measures mixed model with treatment, time and treatment*time interaction term as categorical variables and baseline DAS28 as a continuous variable. A negative change from baseline represents an improvement in assessment of rheumatoid arthritis; LS Mean difference = -0.08, 95% CI 2-sided [-0.397 to 0.240], Standard Error of Mean 0.162 — The direction of comparison is LS mean of GP2013 - LS mean of Rituxan
Statistical Analysis 2: Comparison: MabThera vs GP2013 Part I; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; LS Mean difference = 0.07, 95% CI 2-sided [-0.328 to 0.462], Standard Error of Mean 0.201 — The direction of comparison is LS mean of GP2013 Part I - LS mean of MabThera

5. Secondary Outcome: Number of Patients With ACR20 (CRP) Response
Description: A patient will be considered as improved according the ACR20 criteria
  * at least 20 % improvement from baseline in tender joint count, using the 68-joint count
  * at least 20 % improvement from baseline in swollen joint count, using the 66-joint count
  * and at least 20% improvement from baseline in a least 3 of the following 5 measures:
  * Patient's assessment of RA pain (VAS 100 mm)
  * Patient's global assessment of disease activity (VAS 100 mm)
  * Physician's global assessment of disease activity (VAS 100 mm)
  * Patient self-assessed disability (Health Assessment Questionnaire disability index)
  * Acute phase reactant (C-reactive protein or erythrocyte sedimentation rate)
Time Frame: 24 weeks
Population: PP analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | GP2013 | MabThera | Rituxan | GP2013 Part I
Number analyzed (Participants) | 119 | 76 | 80 | 78
Participants | 86 | 55 | 50 | 56
Statistical Analysis 1: Comparison: GP2013 vs Rituxan; To conclude non-inferiority the lower 95% CI should be greater than -15.0%; Test type: Non-Inferiority — The predefined noninferiority margin of 0.15 for ACR20 is based on the historical placebo-controlled phase III study to evaluate the response rate benefit of adding rituximab to the conventional small molecule-based treatment of patients with RA (Cohen et al. 2006); Response rate difference (%) = 9.77, 95% CI 2-sided [-3.54 to 23.08], Standard Error of Mean 6.79 — The direction of comparison is response rate of GP2013 - response rate of Rituxan
Statistical Analysis 2: Comparison: MabThera vs GP2013 Part I; To conclude non-inferiority the lower 95% CI should be greater than -15.0%; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Response rate difference (%) = -0.57, 95% CI 2-sided [-14.74 to 13.60], Standard Error of Mean 7.23 — The direction of comparison is response rate of GP2013 Part I - response rate of MabThera

6. Secondary Outcome: Summary of Disease Activity According to CDAI
Description: In order to calculate the Clinical Disease Activity Index (CDAI) the number of tender and swollen joints were assessed using the 28 -joint count (tender28 and swollen28). The patient's global assessment of disease activity and the physician's global assessment of disease activity were measured using a Visual Analogue Scale (VAS) of 10 cm (from 0=best to 10=worst).
  CDAI = tender28 + swollen28 + patient's global assessment (in cm) + physician's global assessment (in cm)
Time Frame: At week 24
Population: PP analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | GP2013 | Rituxan | GP2013 Part I | MabThera
Number analyzed (Participants) | 119 | 80 | 78 | 75
Participants
  High disease activity | 26 | 20 | 18 | 18
  Moderate disease activity | 45 | 32 | 24 | 26
  Low disease activity | 41 | 25 | 30 | 19
  Remission | 7 | 3 | 6 | 12

7. Secondary Outcome: Summary of Disease Activity According to SDAI
Description: In order to calculate the Simplified Disease Activity Index (SDAI) the number of tender and swollen joints were assessed using the 28 -joint count (tender28 and swollen28). The patient's global assessment of disease activity and the physician's global assessment of disease activity were measured using a Visual Analogue Scale (VAS) of 10 cm (from 0=best to 10=worst).
  SDAI = CDAI + CRP (in mg/dL)
  (CDAI = tender28 + swollen28 + patient's global assessment (in cm) + physician's global assessment (in cm))
Time Frame: At week 24
Population: PP analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | GP2013 | Rituxan | GP2013 Part I | MabThera
Number analyzed (Participants) | 117 | 77 | 77 | 74
Participants
  High disease activity | 20 | 15 | 13 | 15
  Moderate disease activity | 48 | 34 | 27 | 29
  Low disease activity | 41 | 26 | 31 | 18
  Remission | 8 | 2 | 6 | 12

8. Secondary Outcome: Participant Response as Assessed by EULAR Response Criteria
Description: Present DAS28 ≤ 3.2 (low): good response (if improvement > 1.2), moderate response (if improvement >0.6 and ≤ 1.2), no response (if improvement ≤ 0.6).
  Present DAS28 > 3.2 to ≤ 5.1 (moderate): moderate response (if improvement > 1.2), moderate response (if improvement >0.6 and ≤ 1.2), no response (if improvement ≤ 0.6).
  Present DAS28 > 5.1 (high): moderate response (if improvement > 1.2), no response (if improvement >0.6 and ≤ 1.2), no response (if improvement ≤ 0.6).
Time Frame: At week 24
Population: PP analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | GP2013 | Rituxan | GP2013 Part I | MabThera
Number analyzed (Participants) | 116 | 77 | 76 | 75
Participants
  Good response | 0 | 0 | 0 | 0
  Moderate response | 101 | 61 | 67 | 63
  No response | 15 | 16 | 9 | 12

9. Other Pre Specified Outcome: Number of Patients With at Least One Anti-Drug-Antibody (ADA) Positive Serum Sample
Description: Number of patients with at least one post-baseline Anti-Drug-Antibody (ADA) positive serum sample until the last study visit. Sampling was at Day 1, 29, 113, 169, 267, 365, optional visit 1 (could be at any time between day 169 - week 24 and day 365 - week 52 for patients, who received a 2nd treatment course) and optional visit 2 (only applicable for patients, who received a 2nd treatment course, 26 weeks thereafter, if this was after day 365 - week 52).
Time Frame: through study completion, an average of 1 year
Population: Patients with positive ADA results at randomization were excluded from analysis
Measure: Number; unit: participants
Arm/Group | GP2013 | MabThera | Rituxan
Number analyzed (Participants) | 127 | 84 | 82
participants | 21 | 18 | 11

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) are reported for the entire study duration, which means at least 52 weeks for patients who completed the study. For patients, who received a second optional treatment course, which could be given at any time between week 24 and week 52 an additional follow-up period of 26 weeks after the first infusion of the second treatment course was required. These patients had respectively longer study duration of maximally 1.5 years.
Arm/Group | GP2013 | MabThera | Rituxan
All-Cause Mortality (participants affected / at risk) | 1/133 | 0/87 | 1/92
Serious Adverse Events (participants affected / at risk) | 16/133 | 14/87 | 9/92
Other Adverse Events (participants affected / at risk) | 87/133 | 56/87 | 60/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP2013 (N=133) | MabThera (N=87) | Rituxan (N=92)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — SAEs: Bone marrow failure, Pancytopenia, Sepsis, Septic shock, Multiple organ dysfunction syndrome and Overdose occurred in same patient as a sequence of events due to Methotrexate overdose.
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — SAEs: Bone marrow failure, Pancytopenia, Sepsis, Septic shock, Multiple organ dysfunction syndrome and Overdose occurred in same patient as a sequence of events due to Methotrexate overdose.
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — SAEs chest pain and sinus tachycardia were diagnosed in same patient at the same time
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) — SAEs chest pain and sinus tachycardia were diagnosed in same patient at the same time
Lipogranuloma (General disorders) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) — SAEs: Bone marrow failure, Pancytopenia, Sepsis, Septic shock, Multiple organ dysfunction syndrome and Overdose occurred in same patient as a sequence of events due to Methotrexate overdose.
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — SAEs Fistula, Groin Abscess and Pilonidal cyst occurred in same patient as a sequence of events
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — SAEs Fistula, Groin Abscess and Pilonidal cyst occurred in same patient as a sequence of events
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Purulent pericarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — SAEs: Bone marrow failure, Pancytopenia, Sepsis, Septic shock, Multiple organ dysfunction syndrome and Overdose occurred in same patient as a sequence of events due to Methotrexate overdose.
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — SAEs: Bone marrow failure, Pancytopenia, Sepsis, Septic shock, Multiple organ dysfunction syndrome and Overdose occurred in same patient as a sequence of events due to Methotrexate overdose.
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Bone fissure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — SAEs: Bone fissure, Vitamid D defficiency and Fractured sacrum occurred in same patient as a sequence of events
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — SAEs: Bone fissure, Vitamid D defficiency and Fractured sacrum occurred in same patient as a sequence of events
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — SAEs: Bone marrow failure, Pancytopenia, Sepsis, Septic shock, Multiple organ dysfunction syndrome and Overdose occurred in same patient as a sequence of events due to Methotrexate overdose.
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) — SAEs: Bone fissure, Vitamid D defficiency and Fractured sacrum occurred in same patient as a sequence of events
Fistula (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) — SAEs Fistula, Groin Abscess and Pilonidal cyst occurred in same patient as a sequence of events
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Meningoradiculitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dissociative disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Urogenital prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP2013 (N=133) | MabThera (N=87) | Rituxan (N=92)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 9 (9) | 3 (3) | 5 (10)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 1 (1)
Fatigue (General disorders) | 6 (6) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (3) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 9 (12) | 5 (6) | 9 (11)
Urinary tract infection (Infections and infestations) | 11 (12) | 5 (7) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 6 (7) | 5 (5) | 6 (6)
Bronchitis (Infections and infestations) | 5 (6) | 5 (6) | 1 (1)
Oral herpes (Infections and infestations) | 5 (6) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 5 (5)
Respiratory tract infection (Infections and infestations) | 0 (0) | 3 (4) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 4 (4) | 3 (6) | 2 (2)
Alanine aminotransferase increased (Investigations) | 3 (4) | 1 (1) | 3 (4)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 5 (5)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5) | 8 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (5) | 3 (3)
Headache (Nervous system disorders) | 6 (6) | 5 (7) | 6 (10)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 7 (7)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (5) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 6 (6) | 1 (2)
Hypertension (Vascular disorders) | 5 (5) | 5 (8) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor shall have the right to the first publication or presentation of the results of the study which is intended to be a joint, multi-center publication of the study results. Following the first publication, institutions and/or Principal Investigators may publish or present data or results from the study per the terms of the clinical trial agreement.